| Official Title: | HPV Message Testing and Social Media Campaign |
|-----------------------|-----------------------------------------------|
| NCT number: | 03747302 |
| <b>Document Type:</b> | Survey Information Sheet Phase 2 |
| Date of the | 12/07/2018 |
| <b>Document:</b> | |

# **Information Sheet for Message-Testing Study**

This research project is being conducted by Ardis Olson, MD from the Norris Cotton Cancer Center at Dartmouth and Sunny Kim, PhD from Virginia Commonwealth University. The study is to understand psychological and behavioral effects of messages promoting some pre-teen and teen health topics, including how parents process and respond to those health messages.

You are being asked to take part in a research study about some advertisements because you clicked our [paid ads on social media/Human Intelligence Tasks (HIT's) posted on Amazon Mechanical Turk] for this study. We are interested in your thoughts about health-related messages about pre-teen and teen health. Please read this form carefully and ask any questions you may have before taking part in the study.

**Background:** The purpose of this study is to better understand how people think about different types of health-related messages. This project aims to learn about your psychological reactions and behavioral intentions toward the behavior promoted in the messages.

**Procedures:** If you agree to participate in this study, we will ask you to read a message carefully. You will first be asked a set of questions to determine if you are eligible for the study; these questions are required but you can stop at any time. If you are eligible, you will be asked to complete a survey. We expect this to take less than 15 minutes. You may choose to not answer any or all of these questions. [For MTurk participants only: If you are an MTurk worker, at the end of the survey, you will have to enter your MTurk Worker ID (e.g., XWRTH2WEW345G) and go back to our MTurk HIT to submit the completed task].

## Risks and discomforts

We do not anticipate any risks greater than those encountered in day-to-day life and everyday use of the internet from participating in this research. Please note that the survey is being conducted with the help of Qualtrics, and this software is not affiliated with Dartmouth or Virginia Commonwealth University. It has its own privacy and security policies that you can find at its website.

#### **Benefits**

There are no direct benefits to you.

## Payment for participation

[MTurk workers] You will receive up to 50 cents for finishing the screening question and up to 1.50 cents for taking part in the entire study f. To receive payment, you will have to enter your MTurk Worker ID and go back to our MTurk HIT to submit the completed task. [Participants from social media] You will enter a pool to win one of up to 50 Amazon e-gift cards worth up to \$10 for taking part in the study. To enter the drawing, please click on the link at the end of the survey and provide your contact information. The contact information will be stored separately from your survey responses to protect anonymity of your survey responses.

Voluntary Nature of Participation: Taking part in this study is completely voluntary. You may

skip any questions that you do not want to answer. If you decide not to take part or to skip some of the questions, it will not affect your current or future relationship with Dartmouth College, the Norris Cotton Cancer Center, or Virginia Commonwealth University. If you decide to take part, you are free to withdraw at any time.

Confidentiality: The records of this study, including information collected, will be kept private. Names and other identifying information will not be used in any presentations, papers, or reports written about this project. Your role will be referred to in a generic manner, such as 'Internet users' and 'parents.' Research records will be securely stored in the researchers' offices and on the researchers' password-protected computers. All the digital data (e.g., computer files) will be destroyed (i.e., deleted or erased) when their use is no longer needed but not before a minimum of five years after data collection. Your IP address will be masked from the researchers.

# If you have questions:

Questions about this project can be directed to: Dr. Ardis Olson at the Dartmouth Geisel School of Medicine through the Project Manager, Jenna Schiffelbein. (Jenna.E.Schiffelbein@dartmouth.edu)

If you have any questions or concerns regarding your rights as a subject in this study, you may contact the Institutional Review Board (IRB) at 603-646-6482 or <a href="mailto:CPHS.Tasks@Dartmouth.edu">CPHS.Tasks@Dartmouth.edu</a>, or access their website at <a href="http://www.dartmouth.edu/~cphs/">http://www.dartmouth.edu/~cphs/</a>.

You may print a copy of this form to keep for your records.

Clicking "Next" to begin the study indicates your consent to participate in this study.